CLINICAL TRIAL: NCT04578821
Title: The Effect of Advocacy Education on Developing Social Justice Advocacy Skills and Ethical Sensitivity in Undergraduate Nursing Students: A Randomized Controlled Study
Brief Title: Social Justice Advocacy Skills and Ethical Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nesime Demirören (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor-Investigator, Nesime Demirören, Lecturer, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: t5y4gddx
Record Dates: First submitted 2020-09-10; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Educational Problems
Keywords: patient advocacy; justice; social; nursing education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deney group (Experimental): Education Program:The education program consists of theoretical didactic education, case discussion, film and video screening in class, Web-based laboratory work, SSI practice, poster preparation and awareness activities for a total of 12 weeks and 2 hours per week (24 hours per week).
  Theoretical didactic education, film screening, video screening, Web-based laboratory work, Social Security Institution study, poster preparation, poster presentation at University Campus.
  Interventions: Other: Educational intervention
- Kontrol group (No Intervention): The control group participated in the courses and practices included in the routine curriculum.

INTERVENTIONS:
Other: Educational intervention — Educational intervention
  Arms: Deney group

SUMMARY:
The aim of this study is to determine the effect of advocacy education on social justice advocacy skills and ethical sensitivity in undergraduate nursing students.

DETAILED DESCRIPTION:
Advocacy is an effort to correct or change situations that affect people, society and systems.The origin of advocacy is to provide active support in the Latin "Advocates" dictionary. It is defined as "defense work" in Turkish dictionary advocacy is an ethical dimension of nursing practices in nursing science that shows how nursing care is needed and how the nurse will approach the individual, group and society in need.Social justice advocacy has an increasing importance as people are affected by pressure from the social system.Disease, weakness and early deaths are more common in ethnic and diverse races, poor people and societies that do not receive services.Within the scope of advocacy, the duties and responsibilities of individuals, families and society have been determined by laws and regulations in order to protect and improve the health of the society. Advocacy is the nurse's professional role and ethical responsibility.Total 80 students (İntervention and control group)was selected randomly from 112 4 th grade student. Students were randomly assigned to the experimental group(n=40) and the control group(n=40). The experimental group students will take advocacy intervention courses The control group students will the routine curriculum. In this study, effect size will be determined with 5% error margin by using sample size power analysis Gpower 3.1.9.2 program. Accordingly, it was calculated that 35 students were included in the intervention and control groups with 5% error margin and 80% power. İt was decided to include at least 40 people in each working group with 20% surplus, considering that they might be lost in data collection. Theoretical education, film and video screening, case study, Social Security Institution (SSİ) Study, WEB based work, The student will preparation of advocacy action plan, students prepared poster and advocacy awareness activity, poster were exhibited at the campus. Data Collection Tools: Student Information Form, Social Justice Advocacy Scale , Moral-Ethical Sensitivity Scale. Statistical Analysis:Similarity of experimental and control groups; number, percentage, average and standard deviation, pre-test, post test; scale scores difference in dependent groups t-test.

ELIGIBILITY:
Inclusion Criteria:

* Student who speak very well Turkish

Exclusion Criteria:

* Foreign students who do not speak very well Turkish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Social Justice Advocacy Scale score level | At the beginning of advocacy education, an avarage of 1 hour
  Score level of social justice advocacy skill before advocacy education
Moral Sensitivity Questionnaire score level | At the beginning of advocacy education, an avarage of 1 hour
  Score level of moral sensitivity questionnaire before advocacy education. Similarity of experimental and control groups; number, percentage, average and standard deviation.

SECONDARY OUTCOMES:
Social Justice Advocacy Scale | 12 weeks
  Changes in the score level of social justice advocacy skill after advocacy education
Moral Sensitivity Questionnaire | 12 weeks
  Changes in the score level of moral sensitivity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nesime DEMİRÖREN, Principal Investigator — Selcuk University; Nesime DEMİRÖREN, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol